CLINICAL TRIAL: NCT04653584
Title: Use and Misuse of Domperidone in Parkinson's Disease in France - Observational
Acronym: DUMP-obs
Status: Terminated | Type: Observational
Why Stopped: Administrative problems, the ANSM denied the request to extend the use of the study's budget
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: DUMP-obs
Record Dates: First submitted 2019-02-12; First posted 2020-12-04 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Parkinson Disease patients treated by domperidone according the recommendation
- 2: Parkinson Disease patients treated by domperidone in misuse conditions regarding the recommendation
- 3: Parkinson Disease patients without treathment by domperidone

SUMMARY:
Parkinson disease is the second most frequent neurodegenerative disease after Alzheimer disease and affect 1% of the population over 60 years. The treatment of PD is based on dopamine replacement therapies (DRT). Nausea is the most frequent adverse event whatever the drug, occurring in 30-40% of patients at the initiation of DRT.

Domperidone, a dopamine D2 receptor antagonist with antiemetic properties, does not readily cross the blood-brain barrier, allowing its used in PD. Domperidone may prolong the duration of the QT interval in predisposed patients, and has been associated with proarrhythmia and arrhythmic deaths. Arrhythmias, sudden death and cardiac arrest were reported with high intravenous doses which has led to withdraw of the parenteral form of the drug in 1984. Two case control studies found an increased risk of sudden death associated with domperidone use. In these reports, the increased risk was depending on age, dose, and the use of domperidone in combination with CYP3A4 inhibitors. Following the discussion created by this alert, the PRAC of the EMA has issued recommendations restricting domperidone use to patients younger than 60 years at doses below 30 mg/day and for a short period (7 days).

Because there is no alternative antiemetic drug to be used in PD, domperidone is commonly prescribed as a preventive therapy in most PD patients initiating DRT. In this population, usually older than 60 years, doses of 60 or 80 mg/day are commonly prescribed, for at least 2 months of the DRT escalating dose period or longer. A particular "niche" of domperidone misuse might be patients treated with continuous subcutaneous administration of apomorphine, a second line therapy in PD, inducing severe and prolonged nausea in almost all patients. Little is known about the use of domperidone in PD in France, but misuse of domperidone in PD patients is probably very high. Data collected from two French PD cohorts, COPARK and DIGPD, showed that 8-14% of PD patients were treated with domperidone.

The aim of this proposal is to conduct a cross sectional observational study performed in consecutive patients followed by the 24 PD expert centers of the NS Park network, general hospitals and private practice neurologists, to describe the actual use of domperidone in PD patients.

DETAILED DESCRIPTION:
Domperidone is a dopamine D2 receptor antagonist with antiemetic properties. Domperidone does not readily cross the blood-brain barrier, allowing its used in PD. Domperidone may prolong the duration of the QT interval in predisposed patients, and has been associated with proarrhythmia and arrhythmic deaths. Arrhythmias, sudden death and cardiac arrest were reported with high intravenous doses which has led to withdraw of the parenteral form of the drug in 1984. More recently, two case control studies found an increased risk of sudden death associated with domperidone use. In these reports, the increased risk was depending on age, dose, and the use of domperidone in combination with CYP3A4 inhibitors. Following the discussion created by this alert, the Pharmacovigilance Risk Assessment Committee (PRAC) of the European Medicines Agency (EMA) has issued recommendations restricting domperidone use to patients younger than 60 years at doses below 30 mg/day and for a short period (7 days).

Because there is no alternative antiemetic drug to be used in PD, domperidone is commonly prescribed as a preventive therapy in most PD patients initiating DRT since more than 30 years. In this population, usually older than 60 years, doses of 60 or 80 mg/day are commonly prescribed, for at least 2 months of the DRT escalating dose period or longer. A particular "niche" of domperidone misuse might be patients treated with continuous subcutaneous administration of apomorphine, a second line therapy in PD, inducing severe and prolonged nausea in almost all patients. Little is known about the use of domperidone in PD in France in clinical practice, but misuse of domperidone in PD patients is probably very high. Data collected from two French PD cohorts, COPARK and DIGPD, showed that 8-14% of PD patients were treated with domperidone, extrapolating 10,000 to 20,000 potentially exposed patients at particularly high risk of sudden death.

The aim of this proposal is to conduct a cross sectional observational study of domperidone prescription in PD patients consecutively recruited by neurologists both in University hospitals (24 PD expert centers, thanks to NS-Park/FCRIN network), general hospitals and private neurologists. This will provide insights about the current prescription of domperidone, their doses and duration, the PD patients' profiles, and the different indications for which it is prescribed.

This project will allow describing the use and misuse of domperidone in the PD population in France. This prospective study will take advantage of the recently released national database for PD, supported by the French Plan for Neurodegenerative Disease and by the French Network for Parkinson's disease and Movement Disorders (NS-Park/FCRIN network). This study will help to set up a tool and standardized operating procedures that can be used for subsequent similar studies on clinical practice in neurodegenerative diseases through a large network of academic and private specialists. This information will help Regulatory Authorities to communicate about the safety profile of the drug. Finally, our results obtained in the French population will be compared to those from the European Union countries using domperidone and from which data has been published.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with a diagnosis of Parkinson's disease according to the UKPDSBB criteria and followed-up in consultation or hospitalization in the participating centers

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Parkinson's disease according to the UKPDSBB criteria
Sampling Method: Non-Probability Sample
Enrollment: 1579 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Proportion of Parkinson Disease patients treated by domperidone in misuse conditions regarding the recommendation | Inclusion visit, day 1

SECONDARY OUTCOMES:
Daily dosage of domperidone | Inclusion visit, day 1
Duration of treatment with domperidone | Inclusion visit, day 1
Indications for the prescription of domperidone | Inclusion visit, day 1
Safety measures taken before domperidone prescription in PD patients : ECG (before and after the prescription of domperidone), consultation with a cardiologist and other safety measures | Inclusion visit, day 1
Use of domperidone in combination with contraindicated drugs indicated with domperidone or at risk of contraindicated drug interactions | Inclusion visit, day 1
Presence of medical conditions such as severe hepatic heart failure or cardiac conditions | Inclusion visit, day 1
Symptoms for which domperidone is prescribed | Inclusion visit, day 1

CONTACTS AND LOCATIONS:
Locations (1):
- La Pitié Salpétrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodological sound proposal